CLINICAL TRIAL: NCT01408758
Title: Creating a Virtual Clinician Research Tool
Brief Title: Virtual Clinician Research Tool
Acronym: VCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Geoffrey Williams, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 033339; 5R21DA024262-02 (NIH)
Record Dates: First submitted 2011-01-17; First posted 2011-08-03 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Elevated Risk of Cardiovascular Disease; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VCRT (Other): This group will have 2 visits with a study physician in addition to using the VCRT.
  Interventions: Other: Virtual Clinician Research Tool (VCRT)
- no VCRT (Other): This group will have 2 visits with study physician only, no VCRT.
  Interventions: Other: No VCRT, only physician counseling at visits

INTERVENTIONS:
Other: Virtual Clinician Research Tool (VCRT) — The Virtual Clinician Research Tool (VCRT) will use Self-Determination Theory (SDT) to guide the process or style of how two national guidelines (one for hyperlipidemia, 1 for tobacco dependence)will be operationalized into a virtual format that patients can access online using any internet connected personal computer to develop their plan for change (in this project regarding tobacco or nutrition).
  Arms: VCRT
Other: No VCRT, only physician counseling at visits — No intervention
  Arms: no VCRT

SUMMARY:
The Virtual Clinician Research Tool (VCRT) will use a virtual format to present our National Cholesterol Education Program (Brown, 2004) and the Tobacco Use and Dependence Treatment Clinical Guideline (Fiore et al., 2008) integrated with principles of human motivation from Self-Determination Theory (SDT) for patients with elevated risk for cardiovascular disease from LDL-cholesterol or tobacco dependence.

DETAILED DESCRIPTION:
Hypercholesterolemia and tobacco use interact to increase cardiovascular disease (USDHHS 1990; 2004). Smoking is a cause of metabolic syndrome and diabetes (Eliasson, 2003; Hu et al., 2001; Weitzman et al., 2005). Smokers live on average 13 years less than non-smokers (USDHHS, 2004), and tobacco remains the number one health threat in the United States (Mokdad, Marks, Stroup, & Gerberding, 2004). The Public Health Service (PHS) has published a Guideline for Tobacco Dependence Treatment (Fiore, 2000; Fiore et al., 2008). Hypercholesterolemia is a major risk for cardiovascular disease, and effective treatment with lifestyle and medications lower the risk of cardiovascular events including sudden death, myocardial infarction, and stroke. The National Cholesterol Education Program (NCEP) has published clinical guidelines for its management (Brown, 2004). These include recommendations for therapeutic lifestyle change and medications.

The specific aims of the proposed work are: first, to determine abstinence from tobacco at 6-months and lower LDL-cholesterol from baseline to 6-months for patients assigned the VCRT in addition to the clinician compared to those just receiving clinician care; second, to test for increase in medication use (number of days of medication use-for tobacco dependence mediations and for statin medications for cholesterol) for those receiving the VCRT + clinician; third, to examine the self-determination process model, expanded to include autonomous motivation and perceived competence for medication adherence and actual adherence to promote maintained abstinence and lower LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Tobacco Dependence: Subjects must be currently smoking at least 5 cigarettes per day in the past month, and have smoked 100 cigarettes in their lifetime to qualify for the tobacco VCRT; and will be eligible regardless of their desire to stop smoking.

B. Inclusion Criteria Cholesterol. Subjects must have moderate or moderately high risk for coronary artery disease defined by NCEP (two or more of the following risk factors (male age > 45 years, female >55, HDL-C <40 mg/dl, active smoking, family history of CHD age < 55 years male or age < 65 years female) and the average of two LDL-cholesterols > 100 mg/dl, or the average of two non-HDL cholesterols of 130 mg/dl. Participants will be eligible regardless of desire to lower their cholesterol.

-

Exclusion Criteria:

Exclusion Criteria Tobacco and Cholesterol: Participants will be excluded if they are pregnant or lactating, have a psychotic disorder, are unable to make decisions about medications for themselves, are too sick to participate, or have a life expectancy of less than 12 months (e.g., advanced cancer). Participants will be excluded from the tobacco portion of the trial if they have suicidal ideation (score of 1 or more on the suicidal thought or self harm question in the Patient Health Questionnaire (PHQ) 9). Participants will be excluded from the cholesterol portion of the trial if they have had a heart attack or a stroke, if they have diabetes mellitus, aortic aneurysm, peripheral vascular disease, or chronic kidney disease. They will also be excluded if they are already taking a statin medication to lower their cholesterol. They will be excluded if they are unable to take any of the statin medications due to allergy or adverse reaction in the past (before the study starts). They will be excluded from both cholesterol and tobacco portions of study if they do not speak or write English. Participants will be excluded if they do not have access to a personal computer at home (Mac or PC) with broadband internet access (such as cable modem or digital subscriber line [DSL] and Firefox, Internet Explorer 7 (or higher), or Safari browser software.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tobacco abstinence or lowered LDL cholesterol | 6 months
  abstinence from tobacco at 6-months and lower LDL-cholesterol from baseline to 6-months for patients assigned the VCRT in addition to the clinician compared to those receiving standard clinician care;

SECONDARY OUTCOMES:
increase in medication use | 6 months
  increase in medication use (number of days of medication use-for tobacco dependence mediations and for statin medications for cholesterol) for those receiving the VCRT + clinician;

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C. Williams, M.D., Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center Healthy Living Center, Rochester, New York, United States